CLINICAL TRIAL: NCT04961255
Title: Effects of Post-COVID-19 on Neural Activation and Architecture of the Quadriceps Femoral Muscle-tendon Unit and Its Correlation With Inflammatory Markers
Brief Title: Effects of Post-COVID-19 on Quadriceps Femoral Muscle-tendon Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, João Luiz Q. Durigan, Physical Therapist, Assistant Professor, University of Brasilia
Other Study IDs: CAAE: 45043821.0.0000.8093
Record Dates: First submitted 2021-07-06; First posted 2021-07-14 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Post-COVID-19; Healthy Participants
Keywords: COVID-19; muscle; tendon; cytokines; electrodiagnosis; fatigue; strength; peripheral oxygen extraction
MeSH Terms: conditions — COVID-19; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples to assess cytokines and matrix metalloproteinases (MMPs) involved in COVID-19 pathology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Healthy individuals will be evaluated only once throughout the study. Inflammatory markers, the isometric maximum voluntary force of knee extensor torque, muscle fatigue, neuromuscular adaptations, muscle architecture, quadriceps tendon properties, peripheral oxygen extraction, and body composition will be evaluated.
- COVID-19 positive participants who had moderate symptoms group: These participants will be evaluated 4 times throughout the study.
  Baseline 1: This will be performed between 21 to 30 days after the onset of symptoms of COVID-19 infection.
  Assessment 2: This will be performed between 31 to 90 days after the onset of symptoms of COVID-19 infection.
  Assessment 3: This will be carried out between 91 and 180 days after the onset of symptoms of COVID-19 infection.
  Assessment 4: This will be performed between 181 to 360 days after the onset of symptoms of COVID-19 infection.
  Inflammatory markers, the isometric maximum voluntary force of knee extensor torque, muscle fatigue, neuromuscular adaptations, muscle architecture, quadriceps tendon properties, peripheral oxygen extraction, and body composition will be evaluated in each assessment.
- COVID-19 positive participants who had severe symptoms group: These participants will be evaluated 4 times throughout the study.
  Baseline 1: This will be performed between 21 to 30 days after the onset of symptoms of COVID-19 infection.
  Assessment 2: This will be performed between 31 to 90 days after the onset of symptoms of COVID-19 infection.
  Assessment 3: This will be carried out between 91 and 180 days after the onset of symptoms of COVID-19 infection.
  Assessment 4: This will be performed between 181 to 360 days after the onset of symptoms of COVID-19 infection.
  Inflammatory markers, the isometric maximum voluntary force of knee extensor torque, muscle fatigue, neuromuscular adaptations, muscle architecture, quadriceps tendon properties, peripheral oxygen extraction, and body composition will be evaluated in each assessment.

SUMMARY:
The physiological/biomechanical characteristics related to muscle and tendon architecture and their possible relationship with the loss of muscle strength and fatigue in patients who were infected with COVID-19 are totally unknown. The aim of this study is to evaluate inflammatory markers, the isometric maximum voluntary force of the knee extensor torque, muscle fatigue, neuromuscular adaptations, muscle architecture, tendinous properties of quadriceps components, oxygen extraction, and body composition in participants after diagnosis with Covid-19 who had moderate and severe levels of involvement compared to a healthy control group.

DETAILED DESCRIPTION:
The groups will be composed of participants who had COVID-19, except for the control group, which will be composed of healthy participants who did not have COVID-19. Participants will be divided into: (1) control group, (2) COVID-19 positive participants who had moderate symptoms, (3) COVID-19 positive participants who had severe symptoms. Participants will be recruited from 21 days after the onset of symptoms, the period recommended by the scientific community that the patient no longer transmits severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). After recruitment, 4 evaluations will be carried out over 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Control group:

  - The control group will include healthy participants, aged 18 and 80 years, who had not tested positive for COVID-19.
* COVID-19 positive participants who had moderate symptoms group:

  * Female and male participants, aged between 18 and 80 years, who had Molecular test (RT-PCR) or serological test, which assesses whether the samples are reactive to immunoglobulin M (IgM) and immunoglobulin G (IgG) antibodies, positive for COVID-19;
  * Presence of some of the following symptoms, without the need for hospitalization: dry cough, runny nose, sore throat, diffuse body pain, persistent hyperthermia, no hypoxemia.
* COVID-19 positive participants who had severe symptoms group:

  * Female and male participants, aged between 18 and 80 years, who had Molecular test (RT-PCR) or serological test (which assesses whether the samples are reactive to IgM and IgG antibodies) positive for COVID-19;
  * Presence of hypoxemia (peripheral oxygen saturation - SPO2 ≤ 93%) requiring hospitalization with or without intubation, in addition to the symptoms described for the COVID-19 positive participants who had moderate symptoms group.

Exclusion Criteria:

* Body Mass Index (BMI) ≥ 35 kg/m2;
* Pregnancy;
* Pain, swelling, dermal damage, deformity, or amputation in the regions to be examined;
* Diagnosis of ankylosing spondylitis, rheumatoid arthritis, severe heart disease, advanced chronic obstructive pulmonary disease, cognitive impairment, chemical dependency, psychiatric illness, or behavioral that makes it difficult to cooperate with the procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female and male participants aged between 18 and 80 years who had tested positive for COVID-19 will be included in this study. In addition, the control group will include healthy participants who had not tested positive for COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Blood biomarkers | Change from baseline 1 (days 21-30) to assessments 2 (days 31-90), 3 (days 91-180), and 4 (days 181 to 360) for groups composed of COVID-19 positive participants. The Control group will be assessed only at baseline.
  Blood biomarkers including metalloproteinase 9, interleukin-6, interleukin-8 and interleukin-10, interleukin 1 beta, tumor necrosis factor alpha type, nitric oxide, as well as creatine kinase will be collected in blood samples by venipuncture in the vein brachial, in heparinized tubes with separating gel using the vacutainer system with ethylenediaminetetraacetic acid (EDTA). The samples will be stored and later analyzed using appropriate techniques.
Sit to stand test | Change from baseline 1 (days 21-30) to assessments 2 (days 31-90), 3 (days 91-180), and 4 (days 181 to 360) for groups composed of COVID-19 positive participants. The Control group will be assessed only at baseline.
  To carry out the test will be used a stopwatch and a chair with the back against a wall, seat height 43 cm from the floor and without armrest. The test consists of measuring how many times the participant can get up and sit down from a chair (counting as a movement) in a period of 30 seconds.
Electrodiagnostic stimulus test | Change from baseline 1 (days 21-30) to assessments 2 (days 31-90), 3 (days 91-180), and 4 (days 181 to 360) for groups composed of COVID-19 positive participants. The Control group will be assessed only at baseline.
  The quadriceps femoris, gastrocnemius, soleus and tibialis anterior muscles will be evaluated. At the muscle motor point, the values of rheobase, chronaxia and accommodation will be investigated.
Body composition | Change from baseline 1 (days 21-30) to assessments 2 (days 31-90), 3 (days 91-180), and 4 (days 181 to 360) for groups composed of COVID-19 positive participants. The Control group will be assessed only at baseline.
  Body composition will be estimated using dual x-ray absorptiometry. Fat mass and fat-free mass will be expressed in absolute values.
Muscle force | Change from baseline 1 (days 21-30) to assessments 2 (days 31-90), 3 (days 91-180), and 4 (days 181 to 360) for groups composed of COVID-19 positive participants. The Control group will be assessed only at baseline.
  Muscle force will be assessed by muscle force changes, based on the torque generated during maximum voluntary contraction.
Peripheral oxygen extraction | Change from baseline 1 (days 21-30) to assessments 2 (days 31-90), 3 (days 91-180), and 4 (days 181 to 360) for groups composed of COVID-19 positive participants. The Control group will be assessed only at baseline.
  The assessment of peripheral oxygen extraction will be performed both in rest and during voluntary contraction. The evaluation will be carried out by means of near-infrared spectroscopy (NIRS or near infrared spectroscopy).
Surface electromyographic activity | Change from baseline 1 (days 21-30) to assessments 2 (days 31-90), 3 (days 91-180), and 4 (days 181 to 360) for groups composed of COVID-19 positive participants. The Control group will be assessed only at baseline.
  Electromyographic activity of each superficial component of the quadriceps muscle both in rest and during voluntary contraction.
Muscle architecture | Change from baseline 1 (days 21-30) to assessments 2 (days 31-90), 3 (days 91-180), and 4 (days 181 to 360) for groups composed of COVID-19 positive participants. The Control group will be assessed only at baseline.
  Muscle architecture analyzes will be performed using ultrasound at rest and during voluntary contraction. The muscle volume of the knee extensors, muscle thickness, pennation angle, fascicle length and muscle echogenicity will be evaluated.
Properties of the patellar tendon | Change from baseline 1 (days 21-30) to assessments 2 (days 31-90), 3 (days 91-180), and 4 (days 181 to 360) for groups composed of COVID-19 positive participants. The Control group will be assessed only at baseline.
  The morphological, material and mechanical properties will be evaluated based from the elongation of the patellar tendon during maximum voluntary contraction.
Muscle fatigue | Change from baseline 1 (days 21-30) to assessments 2 (days 31-90), 3 (days 91-180), and 4 (days 181 to 360) for groups composed of COVID-19 positive participants. The Control group will be assessed only at baseline.
  Quadriceps muscle fatigue will be assessed in each leg after consecutive maximal isometric voluntary contractions of the quadriceps muscle.
Assessment of perceived exertion during the fatigue protocol | Change from baseline 1 (days 21-30) to assessments 2 (days 31-90), 3 (days 91-180), and 4 (days 181 to 360) for groups composed of COVID-19 positive participants. The Control group will be assessed only at baseline.
  Assessment of perceived exertion will be analyzed before, during, and after the performance of maximum voluntary isometric contractions performed to analyze muscle fatigue using the BORG scale of perceived exertion.
Fatigue severity analysis | Change from baseline 1 (days 21-30) to assessments 2 (days 31-90), 3 (days 91-180), and 4 (days 181 to 360) for groups composed of COVID-19 positive participants. The Control group will be assessed only at baseline.
  Fatigue severity analysis will be assessed using the fatigue severity scale.

CONTACTS AND LOCATIONS:
Overall Officials: João LQ Durigan, PhD, Principal Investigator — University of Brasilia
Locations (1):
- University of Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Almeida IDS, Ferreira LGJ, Vaz MA, Cipriano Junior G, de Resende MA, Vieira DCL, Costa RR, Babault N, Marqueti RC, Durigan JLQ. Fatigue and neuromuscular function in long COVID: A one-year follow-up study. PLoS One. 2025 Sep 24;20(9):e0332242. doi: 10.1371/journal.pone.0332242. eCollection 2025. PMID 40991619